CLINICAL TRIAL: NCT00183456
Title: Network HIV Prevention Intervention for Drug Users
Brief Title: A Peer-Oriented HIV Prevention Outreach Program for Individuals at High Risk for HIV and Other STIs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH066810 (NIH); R01MH066810 (NIH); DAHBR 9A-ASI
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2012-10-18 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: Sex Education; Peer Group; Social Identity Theory; HIV Seronegativity; Intervention; women; Social Networks; Peer Education
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (4):
- Intervention Condition: CHAT (Experimental): Participants received the program over the course of five small group sessions and one individual session based on a harm reduction philosophy. Participants were trained as Peer Mentors and were encouraged to talk to their family, friends, and sex partners about a range of sex risk reduction options.
  Interventions: Behavioral: Peer-oriented intervention
- Comparison Condition: Standard of Care (Active Comparator): The comparison condition consisted of one group session. The session focused on HIV and STIs transmission and risk reduction information.
  Interventions: Behavioral: Group cognitive behavioral therapy (CBT)
- Network Participants (No Intervention): Index participants generated a list of network members during their baseline visits and were asked to recruit eligible network members into the study. These network participants completed study interviews but did not participate in the intervention.
- Non-randomized Baseline index participants (No Intervention): This arm includes those index participants that did not show up for randomization or did not recruit a network member were thus not eligible to be randomized into a study condition.

INTERVENTIONS:
Behavioral: Peer-oriented intervention — The peer-oriented intervention program emphasized social identity and the goals of protecting family and community. The peer program also trained participants to provide HIV/STD education to their peers.
  Arms: Intervention Condition: CHAT
Behavioral: Group cognitive behavioral therapy (CBT) — Group CBT will focus on teaching ways to modify thoughts and behaviors associated with risky sexual behaviors.
  Arms: Comparison Condition: Standard of Care

SUMMARY:
This study will determine the effectiveness of a peer outreach intervention in preventing HIV infection in adults at high risk for contracting HIV and other sexually transmitted diseases (STDs).

DETAILED DESCRIPTION:
The persistence of HIV and STD epidemics indicates that more effective, sustainable preventive interventions are needed, particularly for low-income, inner-city populations. This study will determine the effectiveness of a theoretically based peer outreach program in preventing HIV and STD transmission among adults in the Baltimore, Maryland area.

Participants will be randomly assigned to receive either a network-oriented peer program emphasizing one's social identity and the goals of protecting one's family and community or group cognitive behavioral therapy (CBT). The peer program will also train participants to provide HIV/STD education to their peers. Participants will be assessed at study entry and during several subsequent follow-up visits. At these study visits, participants will complete questionnaires about their sexual health knowledge and sexual behaviors. Participants and members of their peer network will have follow-up visits at Months 6, 12, and 18.

ELIGIBILITY:
Inclusion Criteria for CBT or Peer Intervention Participants:

1. Female
2. Age 18-55
3. Did not inject drugs in the past 6 months
4. Self-reported sex with at least 1 male partner in the past 6 months
5. Had at least 1 of the following sexual risk factors:

   1. More than 2 sex partners in the past 6 months
   2. STI diagnosis in the past 6 months
   3. Had a high risk sex partner in the past 90 days (i.e. a sex partner that injected drugs, smoked crack, was HIV+, or MSM)

Inclusion Criteria for Peer Network Participants:

1. 18 years old or older
2. One of the following:

   1. Injected drugs
   2. Sex partner of index
   3. Social network member that the index felt comfortable talking to about HIV/STIs

Exclusion Criteria for All Participants:

* Currently enrolled in another HIV prevention intervention

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2005-09; Primary Completion 2007-07 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl A. Latkin, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- The Lighthouse, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The sample consisted of women and their social network members. Index participants were recruited through street outreach as well as at health clinics, and other local community agencies. Social network members were recruited by index participants after completion of the index's baseline visit. Recruitment took place from September 2005-July 2007
Pre-assignment Details: Those index participants that did not recruit a network member or did not show up to be randomized into a study condition were not assigned to a study condition. Network participants completed study interviews but were not assigned to a study condition and did not participate in the intervention.
Period: Overall Study
Arm/Group | Intervention Condition: CHAT | Comparison Condition: Standard of Care | Network Participants | Non-randomized Baseline Index Participants
Started | 85 | 84 | 329 | 248
6 Month Follow-up | 74 | 77 | 278 | 175
12 Month Follow-up | 76 | 74 | 267 | 186
18 Month Follow-up | 80 | 81 | 303 | 207
Completed | 82 (total # of intervention participants that completed any follow-up (6, 12, or 18 month Follow-up)) | 83 (total # of comparison condition participants that completed any follow-up) | 313 (total # of network participants that completed any follow-up) | 220 (total # of non-randomized index participants that completed any follow-up)
Not Completed | 3 | 1 | 16 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Condition: CHAT | Comparison Condition: Standard of Care | Network Participants | Non-randomized Baseline Index Participants | Total
Number analyzed (Participants) | 85 | 84 | 329 | 248 | 746
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 2 | 1 | 3
  Between 18 and 65 years | 85 | 84 | 323 | 247 | 739
  >=65 years | 0 | 0 | 4 | 0 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 42.1 (7) | 43.3 (7) | 42.9 (10) | 40.6 (8) | 42 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 84 | 150 | 248 | 567
  Male | 0 | 0 | 179 | 0 | 179
Region of Enrollment [Number; unit: participants]
  United States | 85 | 84 | 329 | 248 | 746

OUTCOME MEASURES:

1. Primary Outcome: Sex Risk Behaviors: Number of Sex Partners (>=2 Sex Partners)
Description: Number of participants that had 2 or more sex partners in the past 90 days.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Intervention Condition: CHAT | Comparison Condition: Standard of Care | Network Participants | Non-randomized Baseline Index Participants
Number analyzed (Participants) | 73 | 75 | 277 | 174
participants | 17 | 29 | 50 | 53
Statistical Analysis 1: Comparison: Intervention Condition: CHAT vs Comparison Condition: Standard of Care; Test type: Superiority or Other; p < 0.01, Generalized Estimating Equations; Odds Ratio (OR) = 0.28, 95% CI 2-sided [0.13 to 0.63]

2. Secondary Outcome: HIV Communication: Talk to Family About HIV or STIs (Past 6 Months)
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Intervention Condition: CHAT | Comparison Condition: Standard of Care | Network Participants | Non-randomized Baseline Index Participants
Number analyzed (Participants) | 73 | 77 | 277 | 173
participants | 61 | 52 | 155 | 117
Statistical Analysis 1: Comparison: Intervention Condition: CHAT vs Comparison Condition: Standard of Care; Test type: Superiority or Other; p = 0.05, Generalized Estimating Equations; Odds Ratio (OR) = 2.68, 95% CI 2-sided [1.22 to 5.89]

3. Primary Outcome: Sex Risk Behaviors: Unprotected Sex With Non-main Partner (Past 90 Days)
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Intervention Condition: CHAT | Comparison Condition: Standard of Care | Network Participants | Non-randomized Baseline Index Participants
Number analyzed (Participants) | 76 | 74 | 264 | 185
participants | 10 | 22 | 47 | 58
Statistical Analysis 1: Comparison: Intervention Condition: CHAT vs Comparison Condition: Standard of Care; Test type: Superiority or Other; p = 0.05, Generalized Estimating Equations; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.16 to 0.84]

4. Secondary Outcome: HIV Communication: Talk to Family About HIV or STIs (Past 6 Months)
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Intervention Condition: CHAT | Comparison Condition: Standard of Care | Network Participants | Non-randomized Baseline Index Participants
Number analyzed (Participants) | 76 | 74 | 264 | 184
participants | 58 | 39 | 124 | 104
Statistical Analysis 1: Comparison: Intervention Condition: CHAT vs Comparison Condition: Standard of Care; Test type: Superiority or Other; p = 0.01, Generalized Estimating Equations; Odds Ratio (OR) = 2.82, 95% CI 2-sided [1.41 to 5.64]

5. Primary Outcome: Sex Risk Behaviors: Unprotected Anal Sex (Past 90 Days)
Time Frame: 18 month
Measure: Number; unit: participants
Arm/Group | Intervention Condition: CHAT | Comparison Condition: Standard of Care | Network Participants | Non-randomized Baseline Index Participants
Number analyzed (Participants) | 80 | 81 | 299 | 205
participants | 5 | 18 | 43 | 35
Statistical Analysis 1: Comparison: Intervention Condition: CHAT vs Comparison Condition: Standard of Care; Test type: Superiority or Other; p = 0.01, Generalized Estimating Equations; Odds Ratio (OR) = 0.24, 95% CI 2-sided [0.09 to 0.68]

6. Primary Outcome: Sex Risk Behaviors: Unprotected Vaginal Sex (Past 90 Days)
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Intervention Condition: CHAT | Comparison Condition: Standard of Care | Network Participants | Non-randomized Baseline Index Participants
Number analyzed (Participants) | 80 | 81 | 299 | 205
participants | 32 | 49 | 123 | 119
Statistical Analysis 1: Comparison: Intervention Condition: CHAT vs Comparison Condition: Standard of Care; Test type: Superiority or Other; p = 0.05, Generalized Estimating Equations; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.25 to 0.87]

7. Primary Outcome: Sex Risk Behaviors: Unprotected Sex With Main Partner (Past 90 Days)
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Intervention Condition: CHAT | Comparison Condition: Standard of Care | Network Participants | Non-randomized Baseline Index Participants
Number analyzed (Participants) | 80 | 81 | 299 | 205
participants | 30 | 50 | 127 | 113
Statistical Analysis 1: Comparison: Intervention Condition: CHAT vs Comparison Condition: Standard of Care; Test type: Superiority or Other; p = 0.01, Generalized Estimating Equations; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.21 to 0.77]

8. Primary Outcome: Sex Risk Behaviors: Unprotected Sex With a Non-main Partner (Past 90 Days)
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Intervention Condition: CHAT | Comparison Condition: Standard of Care | Network Participants | Non-randomized Baseline Index Participants
Number analyzed (Participants) | 80 | 81 | 299 | 205
participants | 8 | 21 | 47 | 51
Statistical Analysis 1: Comparison: Intervention Condition: CHAT vs Comparison Condition: Standard of Care; Test type: Superiority or Other; p = 0.05, Generalized Estimating Equations; Odds Ratio (OR) = 0.33, 95% CI 2-sided [0.14 to 0.79]

9. Primary Outcome: Sex Risk Behaviors: Any High Risk Sexual Behavior (Past 90 Days)
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Intervention Condition: CHAT | Comparison Condition: Standard of Care | Network Participants | Non-randomized Baseline Index Participants
Number analyzed (Participants) | 80 | 81 | 299 | 205
participants | 51 | 69 | 172 | 151
Statistical Analysis 1: Comparison: Intervention Condition: CHAT vs Comparison Condition: Standard of Care; Test type: Superiority or Other; p = 0.01, Generalized Estimating Equations; Odds Ratio (OR) = 0.30, 95% CI 2-sided [0.14 to 0.64]

10. Secondary Outcome: HIV Communication: Talk to Family About HIV or STIs (Past 6 Months)
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Intervention Condition: CHAT | Comparison Condition: Standard of Care | Network Participants | Non-randomized Baseline Index Participants
Number analyzed (Participants) | 78 | 81 | 291 | 202
participants | 56 | 42 | 141 | 113
Statistical Analysis 1: Comparison: Intervention Condition: CHAT vs Comparison Condition: Standard of Care; Test type: Superiority or Other; p = 0.01, Generalized Estimating Equations; Odds Ratio (OR) = 2.41, 95% CI 2-sided [1.25 to 4.65]

ADVERSE EVENTS:
Arm/Group | Intervention Condition: CHAT | Comparison Condition: Standard of Care | Network Participants | Non-randomized Baseline Index Participants
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/84 | 0/329 | 0/248
Other Adverse Events (participants affected / at risk) | 0/85 | 0/84 | 0/329 | 0/248

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No